CLINICAL TRIAL: NCT02296749
Title: Open Label, Randomized, Two-treatment, Two-period, Two-sequence, Cross Over, Single Dose, Oral Bioequivalence Study of Sirolimus Tablets 2 mg Under Fasting Condition
Brief Title: Bioavailability Study of Sirolimus Tablets 2 mg Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-635/08
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2010-03

CONDITIONS: Healthy
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sirolimus tablets 2 mg (Experimental): Sirolimus tablets 2 mg of Dr. Reddys Laboratories Limited
  Interventions: Drug: Sirolimus
- Rapamune (Active Comparator): Rapamune® 2 mg tablets of Wyeth Laboratories, Philadelphia
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Sirolimus tablets 2 mg
  Other Names: Rapamune

SUMMARY:
This study is to assess the Sirolimus Tablets 2 mg of Dr. Reddy's Laboratories Limited, India and Rapamune® (Sirolimus) tablets 2 mg of Wyeth Laboratories, Philadelphia in healthy, adult,human subjects under Fasting conditions.

DETAILED DESCRIPTION:
Open label, randomized, two-treatment, two-period, two-sequence, cross over, single dose, oral bioequivalence study of Sirolimus tablets 2 mg under Fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

i. Provide written informed consent

ii. Must be healthy, adult, human beings within 18 and 45 years of age (both inclusive) weighing at least 50 kg

iii. Having a body mass index between 18.0 and 24.9 (both inclusive), calculated as weight in Kg/height in m2

iv. Must be of normal health as determined by medical history, physical examination and laboratory investigation performed within 28 days prior to the commencement of the study. (Laboratory values must be within normal limits or considered by the physician / investigator to be of no clinical significance)

v. Female Subjects

* Of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence
* Surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject)

Exclusion Criteria:

i. Incapable of understanding the informed consent

ii. Systolic blood pressure less than 90 mm of 140 mm of Hg

iii. Diastolic blood pressure less than 60 mm of 90 mm of Hg

iv. Oral temperature is below 95.0°F or above 98.6°F

v. Pulse rate below 50/min or above 100/min

vi. History of hypersensitivity or idiosyncratic reaction to investigational drug product or any other related drugs

vii. Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function

viii. Consumption of grapefruit for the past ten days prior to the check-in, in each period

ix. Regular smoker who has a habit of smoking more than nine cigarettes per day and has difficulty in abstaining from smoking during sample collection period

x. Habit of alcoholism and difficulty in abstaining from alcohol during the sample collection period

xi. Difficulty in abstaining from xanthene containing food or beverages (like tea, coffee, chocolates and cola drinks) during the sample collection period

xii. Intake of over the counter (OTC) or prescribed medications and enzyme modifying medication or systemic medication for the last 30 days before dosing

xiii. Clinically significant abnormalities and / or with significant diseases

xiv. Confirmed positive in alcohol screening

xv. Confirmed positive in selected drug of abuse

xvi. Participated in any other clinical investigation using experimental drug/donated blood in past 90 days before the date of start of study

xvii. Confirmed positive in urine pregnancy test

xviii. Female detected to be pregnant, breast feeding or who is likely to become pregnant during the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) | predose (0.00) and 0.25, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.25, 2.50, 2.75, 3.00, 3.25, 3.50, 3.75, 4.00, 4.50, 5.00, 6.00, 8.00, 12.00, 16.00, 24.00, 36.00, 48.00 and 72.00 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Dwarakanath, MBBS, Principal Investigator — Bioserve Clinical Research Pvt Ltd
Locations (1):
- Bioserve Clinical Research Pvt. Ltd, Balanagar, Hyderabad, Andhra Pradesh, India